CLINICAL TRIAL: NCT04097626
Title: The Effects, Perceptions, and Attitudes of Previously Sedentary Individuals Starting an Exercise Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, JeJe Noval, Assistant Professor, Department of Nutrition and Dietitics, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5190325
Record Dates: First submitted 2019-09-17; First posted 2019-09-20 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): This group will receive nutrition education during the first week of the study. This group will perform a minimum of 150 minutes of moderate exercise each week and must be spread out in at least 2 days.
  Interventions: Other: nutrition education
- control (Active Comparator): This group will receive no nutrition education. This group will perform a minimum of 150 minutes of moderate exercise each week and must be spread out in at least 2 days.
  Interventions: Other: no nutrition education

INTERVENTIONS:
Other: nutrition education — The experimental group will receive nutrition education once during the study. It will occur at the beginning of the second week. This will consist of a 30-minute interactive lecture and a 15-minute question-and-answer session. The information covered will be basic nutrition principles for good health and to support regular exercise.
  Arms: experimental
Other: no nutrition education — This group will not receive nutrition education.
  Arms: control

SUMMARY:
To examine whether starting an exercise program with or without education can influence dietary choices in previously sedentary of 20-40 years.

DETAILED DESCRIPTION:
Subjects will complete an InBody test, demographic and physical activity survey, and food-frequency questionnaire via Qualtrics. Also, subjects may participate in a focus group and an individual interview.

A minimum of 150 minutes of moderate exercise required each week and must be spread out in at least 2 days.

Over the course of the study, subjects will complete InBody assessments, Food Frequency Questionnaire (items subjects are eating before, during, and after the investigator's study), and possible focus group questions (open-ended questions about thoughts and perceptions on exercise, nutrition knowledge, and health and nutrition history).

ELIGIBILITY:
Inclusion Criteria:

* Men and Women between 20 and 50 years.
* Previously sedentary for at least 6 months but have been exercising between one week and three months.
* Must be able to perform moderate intensity exercise at least two days per week in at least 30-minute sessions.

Exclusion Criteria:

* Pregnant women (self-reported).
* Currently injured that would prevent subjects from exercising.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-01-28 (Actual)

PRIMARY OUTCOMES:
Body Fat Percentage | change between baseline and visit 5 (six weeks after date of enrollment)
  Body fat percentage will be tested using the InBody 770. This test will take less than 5 minutes to complete. The InBody 770 calculates the measured data using bioelectrical impedance. The testing will be done in the morning around the same time for each participant. Participants will be asked to refrain from eating or drinking that morning to be able to get the most accurate reading.

CONTACTS AND LOCATIONS:
Overall Officials: JeJe Noval, PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States